CLINICAL TRIAL: NCT04838886
Title: The Effect of Telerehabilitation Based Pilates Training on Physical Performance and Quality of Life in Multiple Sclerosis Patients
Brief Title: The Effect of Telerehabilitation Based Pilates Training in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Kader Eldemir, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gazi 2
Record Dates: First submitted 2021-03-30; First posted 2021-04-09 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Pilates; Exercise; Telerehabilitation; Physical performance; Balance; Gait; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Fatigue

STUDY DESIGN:
Intervention Model Description: Intervention and control groups
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The intervention group will be received telerehabilitation-based pilates training three times a week for 6 weeks.
  Interventions: Other: Telerehabilitation-based Pilates Exercise
- Waitlist (No Intervention): The control group will be a wait-list group without any additional specific treatment.

INTERVENTIONS:
Other: Telerehabilitation-based Pilates Exercise — The group that will receive telerehabilitation-based pilates training via telerehabilitation
  Arms: Exercise group

SUMMARY:
Multiple Sclerosis (MS) is a chronic inflammatory disease of the central nervous system characterized by myelin, oligodendrocyte, and axon damage. MS usually begins with attacks due to demyelination of axons in the brain, optic nerve, and spinal cord; over time it develops into a neurodegenerative disease associated with neurotrophic support deficiency and neuronal loss. In MS, various loss of strength, balance, fatigue, cognitive and gait disturbances arise in the central nervous system due to sensory and/or motor neuron degeneration. These disorders affect the quality of life by limiting the individual's activities and participation in their daily lives. Therefore, it is important to treat these disorders in the treatment of MS.

There are various pharmacological treatments and invasive procedures for the management of MS symptoms and one of the most commonly used treatment options is rehabilitation. Clinically-based exercise and rehabilitation are some of the most beneficial rehabilitation strategies in people with MS (PwMS). Clinically-based exercise and rehabilitation have been shown to stabilize or improve many physical symptoms of MS including loss of strength, balance dysfunction, impaired mobility, and fatigue. These benefits have led many practitioners to consider physical exercise as a nonpharmaceutical disease-modifying treatment. However, due to various factors such as mobility disorders, fatigue, and related problems, geographic location, time constraints, transportation difficulties, health insurance coverage, and financial burden, clinical-based exercise may be problematic in some pwMS. To overcome these challenges, approaches to rehabilitation have been developed such as telerehabilitation. The telerehabilitation system provides benefits such as continuity in patient education and rehabilitation, showing progress in rehabilitation, making changes in the treatment program, and saving individuals time and financial expenses. It is also an innovative and potential alternative to face-to-face interventions for treating disease-related disorders in pwMS. In literature, there are many studies examining the effectiveness of telerehabilitation in pwMS. According to these studies, ıt has been shown that telerehabilitation, with its technical facilities, had the potential to make clinical interventions widely accessible and effective for MS, however, telerehabilitation-based interventions could not replace traditional interventions but could perfectly complement. It has been found that telerehabilitation improved balance and postural control in MS patients and had no side effects. However, it was emphasized that the evidence levels of the studies were insufficient for methodological reasons. It has been determined additional studies are needed to investigate examining the effect on walking.

Another clinical-based exercise method is Pilates. Pilates is a "core" stability-based exercise method that includes endurance, flexibility, movement, posture, and respiratory control. Studies have shown that Pilates training can improve balance, mobility, and muscle strength, fatigue in pwMS due to its structure consisting of balance and strengthening exercises. When the literature is reviewed in terms of Telerehabilitation based on Pilates in pwMS, it is seen that there are only two studies. In both studies, pwMS were given 20 minutes of yoga, 20 minutes of Pilates, and 20 minutes of dual-task exercise. However, these studies were in the project phase and the results are still not reported. On the other hand, in both studies, Pilates is given as combined training.

As a result, telerehabilitation is an alternative method to MS treatment. In addition, while there are many clinical-based Pilates studies in the literature, telerehabilitation-based Pilates studies are insufficient. Telerehabilitation-based Pilates training studies are needed. Therefore, the investigators planned this study to investigate the effect of telerehabilitation-based pilates training on physical performance and quality of life in pwMS.

DETAILED DESCRIPTION:
This study is planned as a randomized control trial. Patients will be randomly divided into two groups as intervention and control. The intervention group will be received telerehabilitation-based pilates training three times a week for six weeks. Telerehabilitation-based pilates will be provided via videoconferencing.

The first session will be the introduction session, patients will be informed about basic principles of Pilates and it will be included teaching inward movement of the lower abdominal wall and supine exercises of segmental movements involving trunk muscle recruitment to maintain a neutral posture. Afterward the session, a typical session will be included supine, side-lying, quadruped exercise, sitting on the exercise ball, and standing exercises. Exercises will be included thoracic extension, general abdominal strengthening, core stabilization exercises for the deep abdominal muscles. The difficulty of these exercises will be gradually increased and focused on keeping neutral positions of the spine in different gravity orientations. The control group will be a wait-list group without any additional specific treatment. All assessments will be done before and after the 6-week intervention program or waiting period. The demographic characteristics of the participants initially will be taken and the Expanded Disability Status Scale score of those of MS will be recorded. Primary outcomes are balance, gait, core endurance and power, and muscle strength; secondary outcomes are physical activity, fatigue, and quality of life

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Voluntarily participate in research to accept
* Having a diagnosis of "Multiple Sclerosis" by a specialist physician
* Relapse free in the last 3 mounts
* An Expanded Disability Status Scale (EDSS) score less than or equal to 4

Exclusion Criteria:

* Any cardiovascular, orthopedic, visual, hearing, and perception problems that may affect the results of the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Dynamic Balance- Baseline | Assessment will be conducted before the intervention
  Berg Balance Scale. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. (0 = worst,56 = best)
Dynamic Balance-Post intervention | Assessment will be conducted immediately after the intervention.
  Berg Balance Scale. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. (0 = worst,56 = best)
Static Balance- Baseline | Assessment will be conducted before the intervention.
  Biodex Balance System
Static Balance- Post intervention | Assessment will be conducted immediately after the intervention.
  Biodex Balance System
An individual's confidence in performing activities- Baseline | Assessment will be conducted before the intervention.
  Activities-specific Balance Confidence Scale. Items are rated on a 0% to 100% whole number rating scale. (0 = worst,100 = best)
An individual's confidence in performing activities- Post intervention | Assessment will be conducted immediately after the intervention.
  Activities-specific Balance Confidence Scale. Items are rated on a 0% to 100% whole number rating scale. (0 = worst,100 = best)
Exercise capacity- Baseline | Assessment will be conducted before the intervention.
  Six minute walk test
Exercise capacity- Post intervention | Assessment will be conducted immediately after the intervention.
  Six minute walk test
Gait parameters- Baseline | Assessment will be conducted before the intervention.
  Wearable system (G-Walk)
Gait parameters- Post intervention | Assessment will be conducted immediately after the intervention.
  Wearable system (G-Walk)
Functional mobility- Baseline | Assessment will be conducted before the intervention.
  Timed up go test
Functional mobility- Post intervention | Assessment will be conducted immediately after the intervention.
  Timed up go test
Core endurance- Baseline | Assessment will be conducted before the intervention.
  Mcgill core endurance tests
Core endurance- Post intervention | Assessment will be conducted immediately after the intervention.
  Mcgill core endurance tests
Core strength- Baseline | Assessment will be conducted before the intervention.
  Mcgill core strength tests
Core strength-Post intervention | Assessment will be conducted immediately after the intervention.
  Mcgill core strength tests
Muscle Strength outcomes- Baseline | Assessment will be conducted before the intervention.
  Hand dynamometer (Baseline®, White Plains, New York, US)
Muscle Strength outcomes- Post intervention | Assessment will be conducted immediately after the intervention.
  Hand dynamometer (Baseline®, White Plains, New York, US)

SECONDARY OUTCOMES:
Physical activity level- Baseline | Assessment will be conducted before the intervention.
  international physical activity questionnaire (IPAQ). IPAQ assesses physical activity undertaken across a comprehensive set of domains including leisure time, domestic and gardening (yard) activities, work-related and transport-related activity. The items were structured to provide separate scores on walking; moderate-intensity; and vigorous-intensity activity as well as a combined total score to describe overall level of activity. Computation of the total score requires summation of the duration (in minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activity. (0 Metabolic equivalents (MET) minutes/week= worst, >3000 MET minutes/week= best)
Physical activity level- Post intervention | Assessment will be conducted immediately after the intervention.
  international physical activity questionnaire (IPAQ). IPAQ assesses physical activity undertaken across a comprehensive set of domains including leisure time, domestic and gardening (yard) activities, work-related and transport-related activity. The items were structured to provide separate scores on walking; moderate-intensity; and vigorous-intensity activity as well as a combined total score to describe overall level of activity. Computation of the total score requires summation of the duration (in minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activity. (0 Metabolic equivalents (MET) minutes/week= worst, >3000 MET minutes/week= best)
Fatigue severity- Baseline | Assessment will be conducted before the intervention.
  Fatigue severity scale, A self-report scale is a 9-item scale which measures the severity of fatigue. Answers are scored on a seven point scale where 1 = strongly disagree and 7 = strongly agree. This means the minimum score possible is nine and the highest is 63 (9 = best, 63 = worst)
Fatigue severity- Post intervention | Assessment will be conducted immediately after the intervention.
  Fatigue severity scale, A self-report scale is a 9-item scale which measures the severity of fatigue. Answers are scored on a seven point scale where 1 = strongly disagree and 7 = strongly agree. This means the minimum score possible is nine and the highest is 63 (9 = best, 63 = worst)
Impact of fatigue on activities- Baseline | Assessment will be conducted before the intervention.
  Fatigue impact scale. The FIS was developed to assess the symptom of fatigue as part of an underlying chronic disease or condition. Consisting of 40 items, the instrument evaluates the effect of fatigue on three domains of daily life: cognitive functioning, physical functioning, and psychosocial functioning. Answers are scored on a four point scale where 0 = no problem and 4 = extreme problem. (0 = best, 160 = worst)
Impact of fatigue on activities- Post intervention | Assessment will be conducted immediately after the intervention.
  Fatigue impact scale. The FIS was developed to assess the symptom of fatigue as part of an underlying chronic disease or condition. Consisting of 40 items, the instrument evaluates the effect of fatigue on three domains of daily life: cognitive functioning, physical functioning, and psychosocial functioning. Answers are scored on a four point scale where 0 = no problem and 4 = extreme problem. (0 = best, 160 = worst)
Health related quality of life- Baseline | Assessment will be conducted before the intervention.
  Multiple Sclerosis Quality of Life (MSQOL)-54 scale.. There is no single overall score for the MSQOL-54. Two summary scores -physical health and mental health- can be derived from a weighted combination of scale scores. (0=worst, 100=best)
Health related quality of life- Post intervention- Post intervention | Assessment will be conducted immediately after the intervention.
  Multiple Sclerosis Quality of Life (MSQOL)-54 scale.. There is no single overall score for the MSQOL-54. Two summary scores -physical health and mental health- can be derived from a weighted combination of scale scores. (0=worst, 100=best)

CONTACTS AND LOCATIONS:
Overall Officials: Kader Eldemir, PT, MSc., Study Chair — Research Assistant; Arzu Güçlü-Gündüz, PT, PhD, Study Director — Professor
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data but when the statistical analysis of all data are made, all results will be shared

REFERENCES:
- [Derived] Eldemir K, Guclu-Gunduz A, Eldemir S, Saygili F, Ozkul C, Irkec C. Effects of Pilates-based telerehabilitation on physical performance and quality of life in patients with multiple sclerosis. Disabil Rehabil. 2024 May;46(9):1807-1814. doi: 10.1080/09638288.2023.2205174. Epub 2023 May 6. PMID 37147864
- See also: related info — https://pubmed.ncbi.nlm.nih.gov/?term=Web-based+interventions+in+multiple+sclerosis%3A+the+potential+of+tele-rehabilitation
- See also: related info — https://pubmed.ncbi.nlm.nih.gov/29859267/
- See also: related info — https://pubmed.ncbi.nlm.nih.gov/30744491/